CLINICAL TRIAL: NCT04666675
Title: A Phase 3b Randomized, Placebo-Controlled, Double-Blind Study to Evaluate the Efficacy and Safety of Upadacitinib in Adolescent and Adult Subjects With Moderate to Severe Atopic Dermatitis in Brazil
Brief Title: A Study of Oral Upadacitinib Tablets to Assess Change in Disease State in Participants Aged 12-75 Years With Moderate to Severe Atopic Dermatitis in Brazil
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M20-412
Record Dates: First submitted 2020-12-08; First posted 2020-12-14 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Atopic Dermatitis (AD)
Keywords: Atopic Dermatitis; Upadacitinib; ABT-494; Rinvoq
MeSH Terms: conditions — Dermatitis, Atopic | interventions — upadacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Upadacitinib Dose A (Experimental): Participants will receive Upadacitinib Dose A once daily (QD).
  Interventions: Drug: Upadacitinib
- Upadacitinib Dose B (Experimental): Participants will receive Upadacitinib Dose B QD.
  Interventions: Drug: Upadacitinib
- Placebo for Upadacitinib Followed by Upadacitinib Dose A (Experimental): Participants will receive placebo for Upadacitinib followed by Upadacitinib Dose A QD.
  Interventions: Drug: Upadacitinib; Drug: Placebo for Upadacitinib
- Placebo for Upadacitinib Followed by Upadacitinib Dose B (Experimental): Participants will receive placebo for Upadacitinib followed by Upadacitinib Dose B QD.
  Interventions: Drug: Upadacitinib; Drug: Placebo for Upadacitinib

INTERVENTIONS:
Drug: Upadacitinib — Oral; Tablet
  Other Names: Rinvoq; ABT-494
Drug: Placebo for Upadacitinib — Oral; Tablet
  Arms: Placebo for Upadacitinib Followed by Upadacitinib Dose A; Placebo for Upadacitinib Followed by Upadacitinib Dose B

SUMMARY:
Atopic Dermatitis (AD) is a chronic inflammatory skin disease that is characterized by intense itching, oozing and crusting, redness, skin erosion and dry skin. This study will evaluate how well upadacitinib compared to placebo (no medicine) works to treat participants with moderate to severe AD in Brazil. The study will assess change in disease signs and symptoms.

Upadacitinib is an investigational drug being developed for the treatment of Atopic Dermatitis (AD). This study is "double-blinded", which means that neither the trial participants nor the study doctors will know who will be given which study drug. Study doctors put the participants into 1 of 4 groups called treatment arms. Each group receives a different treatment. Participants with a diagnosis of AD will be enrolled. Around 150 participants will be enrolled in the study in approximately 20 sites in Brazil.

Participants will receive the following for up to 52 weeks:

Participants will receive oral upadacitinib tablets once daily for up to week 52. Participants may also receive oral placebo tablets once daily up to week 16 followed by oral upadacitinib tablets once daily up to week 52.

Arm 1: Upadacitinib Dose A up to week 52. Arm 2: Upadacitinib Dose B up to week 52. Arm 3: Placebo up to week 16 followed by upadacitinib Dose A up to week 52. Arm 4: Placebo up to week 16 followed by upadacitinib Dose B up to week 52.

There may be higher burden for participants in this trial compared to their standard of care. Participants will attend monthly visits during the course of the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, and checking for side effects.

ELIGIBILITY:
Inclusion Criteria:

* Body weight >= 40 kg at the Baseline Visit for participants between >= 12 and < 18 years of age.
* Chronic Atopic Dermatitis (AD) with onset of symptoms at least 3 years prior to Baseline and participant meets Hanifin and Rajka criteria.
* Eczema Area and Severity Index (EASI) score >= 16 at the Screening and Baseline Visits.
* Validated Investigator Global Assessment for AD (vIGA-AD) score ≥ 3 at the Screening and Baseline Visits.
* >= 10% body surface area of AD involvement at the Screening and Baseline Visits.
* Worst Pruritus Numerical Rating Scale (NRS) ≥ 4 at Screening and Baseline Visits.
* Documented history (within 1 year prior to the Screening Visit) of inadequate response (IR) to systemic methotrexate (MTX) and/or cyclosporin A (CsA) or not a candidate for systemic treatment with MTX or CsA as a result of intolerance or medical contraindication.

Exclusion Criteria:

* Prior exposure to any systemic Janus kinase (JAK) inhibitor.
* Prior exposure to dupilumab.
* Must not have used the following AD treatments within the specified timeframe prior to Baseline Visit:

  * Corticosteroids, MTX, CsA, azathioprine. phosphodiesterase type 4 (PDE4)-inhibitors, interferon-γ, and mycophenolate mofetil within 4 weeks.
  * Targeted biologic treatments (refer to within 5 half-lives [if known]) or within 12 weeks, whichever is longer.
  * Phototherapy treatment, laser therapy, tanning booth, or extended sun exposure that could affect disease severity or interfere with disease assessments within 4 weeks.
  * Oral or parenteral traditional medicine within 4 weeks.
  * Moisturizers that contain Topical corticosteroids (TCS), Topical calcineurin inhibitor (TCI)s, or topical Phosphodiesterase type 4 (PDE-4) inhibitors within 7 days.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-12-24 (Estimated); Primary Completion 2021-03-23 (Actual); Study Completion 2021-03-23 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving at least a 75% Reduction in Eczema Area and Severity Index (EASI 75) from Baseline | Baseline to Week 16
  The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of atopic dermatitis (AD).
Number of Participants With Adverse Events (AE) | Up to Week 52
  An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Percentage of Participants Achieving at least a 90% Reduction in Eczema Area and Severity Index (EASI 90) from Baseline | Baseline to Week 16
  The EASI is a validated measure used in clinical practice and clinical trials to assess the severity and extent of AD.

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- See also: This clinical study may be evaluating a usage that is not currently FDA approved. Please see US Prescribing Information for approved uses. — https://www.rxabbvie.com